CLINICAL TRIAL: NCT04344392
Title: Evaluation of Ultrasonography as a Screening Tool for Dysphagia in Patients With Stroke: Correlation With Videofluoroscopic Study
Brief Title: Screening of Dysphagia Via Ultrasonography in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 71306642-050.05.05.04
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Dysphagia, Oropharyngeal; Stroke
Keywords: Hemiplegia; Dysphagia; Ultrasound; Videofluoroscopy
MeSH Terms: conditions — Deglutition Disorders; Stroke; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Single group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to ultrasonographic measurements. Statistical analysis will be performed by an independent consultant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dysphagic hemiplegic patients (Other): Dysphagic patients with hemiplegia as assessed by clinical examination
  Interventions: Diagnostic Test: Ultrasonographic study; Diagnostic Test: Videofluoroscopic study temporal parameters; Diagnostic Test: Videofluoroscopic study distance parameters
- Control (Other): Volunteers which do not have an active swallowing dysfunction.
  Interventions: Diagnostic Test: Ultrasonographic study

INTERVENTIONS:
Diagnostic Test: Ultrasonographic study — Thyroid hyoid approximation and hyoid anterior replacement during swallowing. Tongue thickness in rest.
Diagnostic Test: Videofluoroscopic study temporal parameters — Glossopalatine junction opening and closing time, velopharyngeal junction opening and closing time, laryngeal vestibule opening and closing time, upper esophageal sphincter opening and closing time in seconds.
  Arms: Dysphagic hemiplegic patients
Diagnostic Test: Videofluoroscopic study distance parameters — Hyoid bone horizontal and vertical replacement, thyroid-hyoid approximation (THA) in millimeters.
  Arms: Dysphagic hemiplegic patients

SUMMARY:
Oropharyngeal dysphagia is commonly seen in patients with stroke. Clinical assessment may be used to evaluate dysphagia in patients with stroke however reliability of this method is controversial and videofluoroscopic study is still considered as gold standard. However, exposure to radiation, necessity for a experienced practitioner, an expensive device, and swallowing contrast agents are disadvantages of videofluoroscopy. Ultrasonography, on the other hand, is a cheap, noninvasive device which may demonstrate tongue and laryngeal movement dynamically. In this manner, this study aims to evaluate whether ultrasound can assess dysphagia in patients with hemiplegia accurately.

DETAILED DESCRIPTION:
For a safe swallowing tongue muscles must function properly and larynx should replace superoanterior to close trachea via stretching cricopharyngeal muscle. In this context, approximation of thyroid cartilage and larynx is important for swallowing. These mechanisms are impaired in stroke, Parkinson's disease, traumatic brain injury, and neuromuscular disorders thus resulting oropharyngeal dysphagia. Clinical examination may be used for assessing dysphagia in those patients however reliability of this method is controversial and videofluoroscopic study is considered as gold standard for assessing dysphagia. Ultrasound is used to assess swallowing functions since 1970s however, the studies commonly focused on tongue thickness and functions. Due to advances in technology besides tongue thickness, ultrasonography may practically demonstrate how larynx and thyroid cartilage approximate and hor larynx moves anteriorly. In literature, three methods came to forefront as evaluation methods for dysphagia: 1) approximation of thyroid cartilage and hyoid bone (THA), 2) tongue thickness in rest (TT), and 3) hyoid bone anterior replacement (HAR). In previous studies, the efficiency of THA for assessing dysphagia via videofluoroscopic study has been demonstrated. However other methods have not been evaluated in dysphagic patients with stroke. Ultrasonography, as a cheap, portable and non-invasive method, is a promising for assessing dysphagia in patients with stroke. In this context, this study aims to test the reliability and efficacy of these three methods via ultrasound in dysphagic stroke patients and test the performance of ultrasound compared to videofluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* stroke diagnosis
* aged 18-75
* dysphagia assessed by bedside examination (phase 1: wet voice or cough after drinking 5 ml clear water is positive, phase 2: if phase 1 is negative, inability of drinking 60 ml of water in 2 minutes without coughing or wet voice is positive)

Exclusion Criteria:

* unable to consent due cognitive dysfunction
* unable to cooperate with videofluoroscopic study
* dysphagia before stroke
* rheumatologic or neuromuscular disorder that may cause dysphagia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Glossopalatine junction opening and closing time | through study completion, an average of 1 year
  Opening and closing time of glossopalatine junction after swallowing via videofluoroscopy in seconds.
Velopharyngeal junction opening and closing time | through study completion, an average of 1 year
  Opening and closing time of velopharyngeal junction after swallowing via videofluoroscopy in seconds.
Laryngeal vestibule opening and closing time | through study completion, an average of 1 year
  Opening and closing time of laryngeal vestibule after swallowing via videofluoroscopy in seconds.
Upper esophageal sphincter opening and closing time | through study completion, an average of 1 year
  Opening and closing time of upper esophageal sphincter after swallowing via videofluoroscopy in seconds.
Hyoid horizontal replacement | through study completion, an average of 1 year
  Maximal horizontal replacement of hyoid bone during swallowing via videofluoroscopy in centimeters.
Hyoid vertical replacement | through study completion, an average of 1 year
  Maximal vertical replacement of hyoid bone during swallowing via videofluoroscopy in centimeters.
Thyroid-hyoid approximation | through study completion, an average of 1 year
  Difference of distance between thyroid cartilage and hyoid bone in rest and swallowing in centimeters via ultrasonography.
Tongue thickness | through study completion, an average of 1 year
  Tongue thickness in cm assessed in rest submentally.
Hyoid anterior replacement | through study completion, an average of 1 year
  Distance of hyoid bone replacement between rest position and swallowing in centimeters via ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Volkan Yurdakul, MD, Study Director — Bezmialem University; Delal Öztürk, MD, Principal Investigator — Bezmialem University
Locations (1):
- Bezmialem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YL, Hsieh SF, Chang YC, Chen HC, Wang TG. Ultrasonographic evaluation of hyoid-larynx approximation in dysphagic stroke patients. Ultrasound Med Biol. 2009 Jul;35(7):1103-8. doi: 10.1016/j.ultrasmedbio.2009.02.006. Epub 2009 May 7. PMID 19427098
- [Background] Hsiao MY, Chang YC, Chen WS, Chang HY, Wang TG. Application of ultrasonography in assessing oropharyngeal dysphagia in stroke patients. Ultrasound Med Biol. 2012 Sep;38(9):1522-8. doi: 10.1016/j.ultrasmedbio.2012.04.017. Epub 2012 Jun 12. PMID 22698507
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630